CLINICAL TRIAL: NCT01471145
Title: Feasibility, Mechanism of Action and Potential Side Effects of Extended Release Depot Naltrexone in Opioid Dependent Patients
Brief Title: Depot Naltrexone Mechanism of Action in Heroin Dependent Patients Using fMRI and SPECT
Acronym: XRNT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Alkermes, Inc. (Industry)
Responsible Party: Principal Investigator, Wim van den Brink, Prof. dr. W. van den Brink, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 60-60600-97-301; 2011-001890-15 (EudraCT Number)
Record Dates: First submitted 2011-11-10; First posted 2011-11-15 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Opioid-Related Disorders; Heroin Dependence
Keywords: opioid dependence; heroin dependence; extended release depot naltrexone; functional Magnetic Resonance Imaging; dopamine transporter; Single Photon Emission Computed Tomography
MeSH Terms: conditions — Opioid-Related Disorders; Heroin Dependence | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depot Naltrexone (Experimental)
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — naltrexone for extended-release injectable suspension, 380 mg/vial, every 4 weeks or once a month
  Other Names: Vivitrol

SUMMARY:
The aim of this project is to study brain functions of 20 heroin addicts (compared to brain functions of 20 healthy controls) just before and during a three month extended release naltrexone treatment using functional MRI and dopamine transporter SPECT.

The following hypotheses are tested:

* XRNT modulates the fMRI response to drug cues in predetermined brain regions.
* The expression of striatal transporters (assessed with SPECT) will decrease after a three-month course of extended release naltrexone

DETAILED DESCRIPTION:
Heroin dependence is a quintessential international health problem, with a significant prevalence. Drug free treatments, including pharmacologically supported interventions using oral naltrexone, have not been very successful, mainly due to low compliance. The recent introduction of Vivitrol®, consisting of monthly injections, may create new opportunities. Vivitrol® is an innovative treatment delivery method that blocks the rewarding effects of heroin.

ELIGIBILITY:
Inclusion Criteria:

* Heroin dependent patients: have a diagnosis of opioid dependence according to DSM-IV criteria, heroin as primary drug of abuse and inhalation as primary route of administration.
* Healthy controls: no diagnosis of substance dependence, no current psychotropic medication. Care will be taken to match controls for gender, age, smoking status, IQ and handedness.

Exclusion Criteria:

* Age below 18 or over 55
* Medical contraindications for XRNT or MRI (Langleben 2006; Langleben, Ruparel et al. 2008). Briefly, the former include candidates with known hypersensitivity to naltrexone,PLG (poly-lactide-coglycolide), carboxymethylcellulose, or any other components of the Vivitrol® diluent, hepatic or renal disease, chronic pain syndromes, female subjects who are pregnant or lactating, or are of child bearing potential and are not using an acceptable method of birth control. MRI contraindications include chronic medical (neurological, cardiovascular, infectious, metabolic, etc) conditions that may affect the brain morphology and/or activity and indwelling foreign metallic or magnetically sensitive objects and devices, such as shrapnel, pacemakers, orthopaedic fixation devices or vascular stents
* Presence of disorders precluding normal perception of visual and auditory stimuli, such as color blindness, deafness, severe myopia, etc.
* Patients with a history of or current psychosis or current major depressive disorder with suicidal ideation
* Patients who are being treated under forced treatment conditions
* History or evidence of disorders that may affect cerebral function or circulation, such as diabetes and other metabolic disorders, encephalopathy, cardiovascular or cerebrovascular disease, history of head trauma with depressed skull fracture or prolonged loss of consciousness and history of brain surgery
* Female subjects: women who are pregnant or breast-feeding
* Current psychotropic medication
* Use of any prescription medications that could affect alertness or the circulatory system
* IQ < 70
* Naltrexone use within the past 6 months
* Baseline aspartate aminotransferase or alanine aminotransferase more than three times the upper limit of normal
* Patients with no intention to be opioid-free for a minimum of 7 days before starting XRNT treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Brain functions | 3 months
  Brain functions of 20 heroin addicts just before and during a three month extended release naltrexone treatment using both functional MRI and dopamine transporter SPECT, compared to brain functions of 20 healthy controls.

SECONDARY OUTCOMES:
Feasibility and potential efficacy | 3 months
  The feasibility and potential efficacy of extended release naltrexone in a pilot sample of 20 Dutch heroin addicts in terms of (a) the percentage of patients that actually starts treatment when invited and (b) the percentage of 3 months retention.

CONTACTS AND LOCATIONS:
Overall Officials: Wim van den Brink, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Background] Cornish JW, Metzger D, Woody GE, Wilson D, McLellan AT, Vandergrift B, O'Brien CP. Naltrexone pharmacotherapy for opioid dependent federal probationers. J Subst Abuse Treat. 1997 Nov-Dec;14(6):529-34. doi: 10.1016/s0740-5472(97)00020-2. PMID 9437624
- [Background] de Geus EJ, van't Ent D, Wolfensberger SP, Heutink P, Hoogendijk WJ, Boomsma DI, Veltman DJ. Intrapair differences in hippocampal volume in monozygotic twins discordant for the risk for anxiety and depression. Biol Psychiatry. 2007 May 1;61(9):1062-71. doi: 10.1016/j.biopsych.2006.07.026. Epub 2006 Nov 29. PMID 17137562
- [Background] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899
- [Background] Krupitsky E, Nunes EV, Ling W, Illeperuma A, Gastfriend DR, Silverman BL. Injectable extended-release naltrexone for opioid dependence: a double-blind, placebo-controlled, multicentre randomised trial. Lancet. 2011 Apr 30;377(9776):1506-13. doi: 10.1016/S0140-6736(11)60358-9. PMID 21529928
- [Background] Langleben DD, Ruparel K, Elman I, Busch-Winokur S, Pratiwadi R, Loughead J, O'Brien CP, Childress AR. Acute effect of methadone maintenance dose on brain FMRI response to heroin-related cues. Am J Psychiatry. 2008 Mar;165(3):390-4. doi: 10.1176/appi.ajp.2007.07010070. Epub 2007 Dec 3. PMID 18056224
- [Background] Lobmaier P, Kornor H, Kunoe N, Bjorndal A. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD006140. doi: 10.1002/14651858.CD006140.pub2. PMID 18425938
- [Background] Luijten M, Veltman DJ, van den Brink W, Hester R, Field M, Smits M, Franken IH. Neurobiological substrate of smoking-related attentional bias. Neuroimage. 2011 Feb 1;54(3):2374-81. doi: 10.1016/j.neuroimage.2010.09.064. Epub 2010 Oct 13. PMID 20932921
- [Background] Suh JJ, Langleben DD, Ehrman RN, Hakun JG, Wang Z, Li Y, Busch SI, O'Brien CP, Childress AR. Low prefrontal perfusion linked to depression symptoms in methadone-maintained opiate-dependent patients. Drug Alcohol Depend. 2009 Jan 1;99(1-3):11-7. doi: 10.1016/j.drugalcdep.2008.06.007. Epub 2008 Jul 31. PMID 18674871
- [Background] Suh JJ, Pettinati HM, Kampman KM, O'Brien CP. Gender differences in predictors of treatment attrition with high dose naltrexone in cocaine and alcohol dependence. Am J Addict. 2008 Nov-Dec;17(6):463-8. doi: 10.1080/10550490802409074. PMID 19034737
- [Background] Zijlstra F, Booij J, van den Brink W, Franken IH. Striatal dopamine D2 receptor binding and dopamine release during cue-elicited craving in recently abstinent opiate-dependent males. Eur Neuropsychopharmacol. 2008 Apr;18(4):262-70. doi: 10.1016/j.euroneuro.2007.11.002. PMID 18077142
- [Background] Zijlstra F, Veltman DJ, Booij J, van den Brink W, Franken IH. Neurobiological substrates of cue-elicited craving and anhedonia in recently abstinent opioid-dependent males. Drug Alcohol Depend. 2009 Jan 1;99(1-3):183-92. doi: 10.1016/j.drugalcdep.2008.07.012. Epub 2008 Sep 26. PMID 18823721